CLINICAL TRIAL: NCT05629572
Title: Clinical Evaluation of the i-STAT High Sensitivity Troponin I Test to Aid in the Diagnosis of Myocardial Infarction (MI)
Brief Title: Abbott i-STAT High Sensitivity Troponin I Study
Acronym: i-STAT hs-TnI
Status: Completed | Type: Observational
Sponsor: Abbott Point of Care (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-2020-0012
Record Dates: First submitted 2022-11-11; First posted 2022-11-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lithium Heparin (LiH) plasma stored in cryovial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Prospective subjects in Emergency Department (ED) with symptoms of acute coronary syndrome (ACS).: Prospectively collected whole blood specimens from subjects presenting to the emergency department (ED) with chest discomfort or equivalent ischemic symptoms suggestive of acute coronary syndrome (ACS).
  For this study's MI adjudication, a minimum of 2 samples are to be tested on the site's standard of care (SOC) instrument, one at baseline and one at another time point (T1, T2, T3). For each of the SOC test results, a corresponding research draw for testing on the i-STAT hs-TnI cartridge should be attempted, if feasible. For research, a minimum of 2 samples are to be tested on i-STAT instruments, one at baseline and one at an additional timepoint. Enrollment will be monitored throughout the clinical study.
  Interventions: Diagnostic Test: i-STAT hs-TnI Cartridge Testing on i-STAT 1 and i-STAT Alinity

INTERVENTIONS:
Diagnostic Test: i-STAT hs-TnI Cartridge Testing on i-STAT 1 and i-STAT Alinity — Paired whole blood and plasma samples collected at multiple time points.

SUMMARY:
The goal of this observational multi-center study is to evaluate the clinical performance of the i-STAT hs-TnI test (i-STAT High Sensitivity Troponin I) using the investigational i-STAT hs-TnI cartridge for the proposed intended use as an aid in the diagnosis and treatment of myocardial infarction (MI). The cartridge measures cardiac troponin I (cTnI) in whole blood or plasma samples using the i-STAT 1 Analyzer or i-STAT Alinity Instrument. Subjects presenting to the emergency department (ED) with chest discomfort or equivalent ischemic symptoms suggestive of Acute Coronary Syndrome (ACS) who are enrolled in this study will be asked to provide blood samples for testing.

DETAILED DESCRIPTION:
The i-STAT High Sensitivity Troponin I (i-STAT hs-TnI) test is an in vitro diagnostic test for the quantitative measurement of cardiac troponin I (cTnI) in whole blood or plasma samples using the i-STAT 1 Analyzer or i-STAT Alinity Instrument in point of care or clinical laboratory settings. The hs-TnI test is intended to be used as an aid in the diagnosis of myocardial infarction (MI).

The objective of this study is to evaluate the clinical performance of the i-STAT hs-TnI test using the investigational i-STAT hs-TnI Cartridge with the i-STAT 1 Analyzer and i-STAT Alinity Instrument for subjects presenting to the emergency department (ED) with chest discomfort or equivalent ischemic symptoms suggestive of acute coronary syndrome (ACS).

The clinical evaluation will use prospectively collected whole blood specimens from subjects presenting to the ED with chest discomfort or equivalent ischemic symptoms suggestive of ACS.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Presenting to the Emergency Department (ED) with signs and symptoms suggestive of Acute Coronary Syndrome (ACS): Acute chest, epigastric, neck, jaw or arm pain or discomfort or pressure without apparent non-cardiac source; Shortness of breath, nausea, vomiting, fatigue/malaise; Other equivalent discomfort suggestive of a myocardial infarction (MI) in accordance with the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines.
* Electrocardiogram (ECG) ordered as part of the standard of care

Exclusion Criteria:

* Previously enrolled in the study
* Enrolled in any interventional clinical trial (within the last 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consisted of subjects presenting to emergency departments (ED) with chest discomfort or equivalent ischemic symptoms suggestive of acute coronary syndrome (ACS) and had an electrocardiogram (ECG) ordered as part of their standard of care (SOC).
Sampling Method: Probability Sample
Enrollment: 3697 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Performance of i-STAT hs-TnI cartridge | Up to 9 hours
  Performance metrics calculated using adjudicated outcomes with the hs-TnI test results.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Gupta, MS, MBA, Study Director — Abbott Point of Care
Locations (28):
- United States (28):
  - Mercy Gilbert Medical Center, Chandler, Arizona
  - University of California at San Francisco, San Francisco, California
  - Stanford Medical Center, Stanford, California
  - Geroge Washington University, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kentucky Clinical Trials Labatory, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin Healthcare (Research Institute/Minneapolis Medical Research Foundation), Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cooper University Hospital, Camden, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Stony Brook University, Stony Brook, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Penn State University Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Florence Medical Centre (MUSC Health), Florence, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Baylor Scott and White Healthcare, Temple, Texas
  - University of Virginia, Charlottesville, Virginia
  - Eastside Research Associates, Redmond, Washington

REFERENCES:
- [Background] Bertrand ME, Simoons ML, Fox KA, Wallentin LC, Hamm CW, McFadden E, de Feyter PJ, Specchia G, Ruzyllo W. Management of acute coronary syndromes: acute coronary syndromes without persistent ST segment elevation; recommendations of the Task Force of the European Society of Cardiology. Eur Heart J. 2000 Sep;21(17):1406-32. doi: 10.1053/euhj.2000.2301. No abstract available. PMID 10952834
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Alpert JS, Eagle KA, Faxon DP, Fuster V, Gardner TJ, Gregoratos G, Russell RO, Smith SC Jr. ACC/AHA guidelines for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on the Management of Patients With Unstable Angina). J Am Coll Cardiol. 2000 Sep;36(3):970-1062. doi: 10.1016/s0735-1097(00)00889-5. No abstract available. PMID 10987629
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Sharma S, Jackson PG, Makan J. Cardiac troponins. J Clin Pathol. 2004 Oct;57(10):1025-6. doi: 10.1136/jcp.2003.015420. No abstract available. PMID 15452153
- [Background] Alushi B, Jost-Brinkmann F, Kastrati A, Cassese S, Fusaro M, Stangl K, Landmesser U, Thiele H, Lauten A. High-Sensitivity Cardiac Troponin T in Patients with Severe Chronic Kidney Disease and Suspected Acute Coronary Syndrome. J Clin Med. 2021 Sep 17;10(18):4216. doi: 10.3390/jcm10184216. PMID 34575325
- [Derived] Wu AHB, Mahler SA, House SL, Jortani SA, Creer MH, Rising KL, Bischof JJ, Crystal C, Headden GF, Apple FS, Harrison NE, Meltzer AC, Baca JT, Tiffany B, Sochor M, Pentecostes GU, Di Tullio KP, Gupta MS, Singer AJ, Januzzi JL. Clinical Performance of a Novel Point-of-Care High-Sensitivity Cardiac Troponin I Assay. J Appl Lab Med. 2026 Jan 5;11(1):98-112. doi: 10.1093/jalm/jfaf152. PMID 41146629